CLINICAL TRIAL: NCT02628080
Title: Pre-operative Window of Opportunity Study of the Effects of Atovaquone on Hypoxia in Non-small Cell Lung Carcinoma
Brief Title: Atovaquone as Tumour HypOxia Modifier
Acronym: ATOM
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OCTO-073
Record Dates: First submitted 2015-09-07; First posted 2015-12-11 (Estimated); Last update posted 2019-09-04 (Actual); Status verified 2019-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Hypoxia
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Hypoxia | interventions — Atovaquone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (Experimental): Atovaquone suspension, 750mg/5ml bd and 1000mg (6.25ml) bd for 7-17 days. Device: PET-CT, Device: DWI-MRI
  Interventions: Drug: Atovaquone
- Cohort 2 (No Intervention): Device: PET-CT, Device: DWI-MRI

INTERVENTIONS:
Drug: Atovaquone — Atovaquone has an EU marketing authorisation (held by Glaxo Wellcome UK Ltd) and is indicated for acute treatment of mild to moderate Pneumocystis pneumonia (PCP). It is also used in combination with proguanil for malaria prophylaxis.
  Other Names: Wellvone
  Arms: Cohort 1

SUMMARY:
Solid tumours often have highly disorganised vasculature that results in low oxygenation. This combined with high metabolic rates leads to oxygen demand outstripping supply causing tumour hypoxia. Hypoxia drives multiple cellular processes involved in the hallmarks of cancer. Tumour hypoxia also decreases the effectiveness of anticancer treatments. This is especially true for patients treated with radiotherapy since it has been long recognised that hypoxic tumour cells require 3 times the dose of radiation to cause the same amount of cell death as cells irradiated under normal oxygen conditions.

To date, the majority of attempts at overcoming tumour hypoxia have focused on increasing oxygen supply. However, such techniques have produced modest benefits at best and subsequently have not been adopted into current clinical practice.

An interesting alternative approach to tackling tumour hypoxia is to decrease oxygen 'demand' by reducing tumour oxygen consumption. This strategy has been suggested to be more effective in reducing hypoxia than previous methods aimed at increasing oxygen delivery.

Pre-clinical data demonstrates that the commonly prescribed anti-protozoal drug atovaquone significantly reduces oxygen consumption in a variety of tumour cell lines in vitro. This reduction in oxygen consumption leads to a profound reduction in tumour hypoxia in animal models. It is anticipated that if these effects on tumour hypoxia could be reproduced in humans, that their tumours could be rendered markedly more sensitive to radiotherapy.

This window of opportunity trial will assess whether atovaquone significantly reduces tumour hypoxia in adult patients referred for surgery with suspected non-small cell lung cancer. This will be assessed using a combination of functional imaging and circulating markers of hypoxia. If atovaquone is demonstrated to result in a reduction in tumour hypoxia, larger clinical trials will be conducted to determine whether this well-tolerated and inexpensive agent improves radiotherapy efficacy and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Suspected NSCLC considered suitable for surgical resection by the lung multidisciplinary team meeting (MDT).
2. At least one measurable lesion (greater than 2.5cm maximal length in any direction) that the investigators consider on routine imaging (CT or PET-CT scan performed in the 60 days prior to consent (older scans may be accepted at the discretion of the Chief Investigator providing the results remain clinically significant)) likely to contain regions of hypoxia.
3. Male or female, Age ≥ 18 years.
4. Eastern Cooperative Oncology Group (ECOG) performance score of 0-2
5. The patient is willing and able to comply with the protocol, scheduled follow-up visits and examinations for the duration of the study.
6. Written (signed and dated) informed consent.
7. Haematological and biochemical indices within given ranges

Exclusion Criteria:

1. Previous systemic chemotherapy or biological therapy within 21 days of commencing atovaquone treatment.
2. Treatment with any other investigational agent, or participation in another interventional clinical trial within 28 days prior to enrolment.
3. Known previous adverse reaction to atovaquone or its excipients.
4. Active hepatitis, gallbladder disease or pancreatitis
5. Patients with impaired gastrointestinal (GI) function or GI disease that may significantly alter absorption of atovaquone.
6. Concurrent administration of contraindicated agents in the 14 days prior to starting atovaquone as outlined in section 9.4 and the current atovaquone Summary of Product Characteristics (SmPC).
7. Concurrent administration of warfarin in the 14 days prior to starting atovaquone.
8. Patients taking known inhibitors of the electron transport chain such as Metformin.
9. Other psychological, social or medical condition, physical examination finding or a laboratory abnormality that the Investigator considers would make the patient a poor trial candidate or could interfere with protocol compliance or the interpretation of trial results.
10. Patients who are known to be serologically positive for Hepatitis B, Hepatitis C or HIV (Hepatitis and HIV testing specifically for confirming eligibility for this trial are not required).
11. Pregnant or breast-feeding women or women of childbearing potential unless highly effective methods of contraception are used.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Percentage change in reduction of hypoxia by atovaquone | Day 0 v Day 7-17, and Day 0 post surgery (tumour sample)
  Average hypoxic volume reduction (%) in 18F-fluoromisonidazole (18F-MISO)/18F-fluoroazomycin arabinoside (18F-FAZA) uptake as detected by hypoxia-PET(positron emission tomography)-CT scans.

SECONDARY OUTCOMES:
Reduction of perfusion by atovaquone | Day 0 v Day 7-17
  Changes in tumour blood flow measured by perfusion CT, DWI-MRI, DCE-MRI and PET kinetic modelling
Replacement of hyp-PET-CT imaging with serological markers of hypoxia | Day 0 v Day 7-17
  Changes in hypoxia-PET-CT derived hypoxic volumes compared with changes in plasma levels of serological markers of hypoxia
Reproducibility | Day 0 v Day 7-17
  Comparison of hypoxia-PET-CT, perfusion CT, serological tests, diffusion-weighted imaging (DWI-MRI) and Dynamic contrast-enhanced MRI (DCE-MRI) derived parameters

OTHER OUTCOMES:
Correlation of hypoxia modification with PK (pharmacokinetic) levels of atovaquone (plasma and tumour) | Day 0 v Day 7-17 for plasma level. Day 0 v Post resection for tumour sample (cohort 1 only)
  HPLC (high pressure liquid chromatography) based measurement of plasma level and tumour level of atovaquone
Correlations between imaging and histology | Day 0 v Day 7-17
  Comparison of histological hypoxia and vasculature parameters with prior imaging measuring hypoxia, perfusion, and glycolysis
Correlations between serological hypoxia markers and histology | Day 0 v Day 7-17
  Comparison of serological hypoxia parameters with immunohistochemistry on pimonidazole staining
To assess whether atovaquone results in a lower level of hypoxia metagene signature expression | Day 0 v Day 7-17
  Hypoxia metagene signature expression and Individual tests to measure gene expression/mutation
Progression-free survival and overall survival | At 12 and 24 months
  Progression-free survival and overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Geoff Higgins, MBChB, MRCP, FRCR, Principal Investigator — University of Oxford
Locations (1):
- Churchill Hospital, Oxford, Oxfordshire, United Kingdom

REFERENCES:
- [Derived] Bourigault P, Skwarski M, Macpherson RE, Higgins GS, McGowan DR. Timing of hypoxia PET/CT imaging after 18F-fluoromisonidazole injection in non-small cell lung cancer patients. Sci Rep. 2022 Dec 16;12(1):21746. doi: 10.1038/s41598-022-26199-7. PMID 36526815
- [Derived] Bourigault P, Skwarski M, Macpherson RE, Higgins GS, McGowan DR. Investigation of atovaquone-induced spatial changes in tumour hypoxia assessed by hypoxia PET/CT in non-small cell lung cancer patients. EJNMMI Res. 2021 Dec 29;11(1):130. doi: 10.1186/s13550-021-00871-x. PMID 34964932